CLINICAL TRIAL: NCT04618484
Title: Can Non-pharmacological BIOmodulation Improve Healing After Arthroscopic Rotator Cuff Repair Using a Knotted Suturebridge Technique?
Brief Title: Biomodulating Rotator Cuff Healing - A Proof of Concept Trial
Acronym: BIOHACK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinique Générale dAnnecy (Other)
Responsible Party: Principal Investigator, Geert Alexander Buijze, Orthopaedic Surgeon, Clinique Générale dAnnecy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020BIOHACK-trial
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biomodulation (Experimental): 6-weeks post-operative cryo-, photo- and electro-biomodulation protocol after repair
  Interventions: Other: Biomodulation (non-pharmacological)
- Control (No Intervention): standard rehabilitation after repair

INTERVENTIONS:
Other: Biomodulation (non-pharmacological) — cryo-, photo- and electro-biomodulation
  Arms: Biomodulation

SUMMARY:
Novel concepts in quantum biology of rotator cuff repair and author's novel findings on biomodulation inspired us to design a pragmatic non-pharmacological add-on rehabilitation protocol that may potentially decrease retear rates after arthroscopic repair using a knotted suturebridge technique. In this proof-of-concept trial, 146 patients will be randomized 1:1 to either a 6-weeks post-operative cryo-, photo- and electro-biomodulation protocol or a control group immobilized in a standard abduction sling for 6 weeks. Healing will be evaluated using the Sugaya classification on MRI at 1 year post-operatively.

ELIGIBILITY:
Inclusion criteria

* Patient is over 18 years old
* Patient presents with a symptomatic full-thickness tear as diagnosed preoperatively on ultrasound, arthro-CT or MRI.
* Absence of significant muscle atrophy or fatty infiltration of the affected tendon exceeding stage 2 of the Goutallier classification

Exclusion criteria

* Partial rotator cuff tear or other shoulder injury
* Planned concomitant procedures other than subacromial decompression, acromioclavicular joint resection or biceps tenodesis/tenotomy
* Irreparable rotator cuff tear
* Patients who present with cartilage lesions greater than stage II of the Outerbridge classification (≥15mm diameter) on preoperative x-ray
* Patient presenting with a known comorbidity that could affect the outcome of surgery (cervical radiculopathy, polyarthritis, neurological disease of the upper limb)
* Patient not able to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Healing of rotator cuff tear | 1 year post-operatively
  Healing will be evaluated using the Sugaya classification on MRI

SECONDARY OUTCOMES:
Patient reported outcome measures | 6 months and 1 year
  Pain, reported as average of reported pain during movement, at rest and at night, measured by a numeric rating scale from 0 to 10; and the Auto-Constant score, Subjective Shoulder Value, the American Shoulder and Elbow Surgeon score Surgeon score
Active range of motion | 6 months and 1 year
  Degrees of forward flexion, abduction, internal rotation and external rotation (90 degrees elbow flexion, 0 and 90 degrees abduction)
Compliance | First 6 weeks after surgery
  Self-reported daily compliance to the different components of the biomodulation protocol
Postoperative complications | First year after surgery
  Postoperative complications in the first year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Générale d'Annecy, Annecy, France

IPD SHARING:
Plan to Share IPD: No
Due to privacy reasons individual patient data will not be available to the public.

REFERENCES:
- [Derived] Allaart LJH, Lech J, Macken AA, Kling A, Lafosse L, Lafosse T, van den Bekerom MPJ, Buijze GA. Biomodulating healing after arthroscopic rotator cuff repair: the protocol of a randomised proof of concept trial (BIOHACK). BMJ Open. 2023 Aug 16;13(8):e071078. doi: 10.1136/bmjopen-2022-071078. PMID 37586862